CLINICAL TRIAL: NCT04438265
Title: Quadratus Lumborum Type 2 as Chronic Hip Pain Treatment
Status: Completed | Type: Observational
Sponsor: Hospital Medina del Campo (Other)
Collaborators: Hospital Universitaio Getafe (Unknown); Hospital Rio Hortega (Unknown)
Responsible Party: Principal Investigator, María Teresa Fernandez, Principal Investigator, Hospital del Rio Hortega
Other Study IDs: PI20-1770 A.4.2/PI 21-PI104
Record Dates: First submitted 2020-06-10; First posted 2020-06-18 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Hip Arthropathy; Chronic Hip Pain; Ultrasound Therapy; Complications
Keywords: chronic hip pain; ultrasound therapy
MeSH Terms: interventions — Levobupivacaine; Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- quadratus lumborum: analgesic technique. The evaluation of the patient will consist of 2 stages. The first of these will consist of the evaluation consultation (clinical history, EVN evaluation, WOMAC) and initial treatment (QL2 block). In the second stage, the patient will be followed up with interviews at 3 weeks, 3 and 6 months.
  Interventions: Drug: levobupivacaine; Device: ultrasound device
- Control: Current analgesia , no QL block apply

INTERVENTIONS:
Drug: levobupivacaine — local anesthetic
  Other Names: chirocane
  Groups: quadratus lumborum
Device: ultrasound device — scream
  Groups: quadratus lumborum

SUMMARY:
The main objective of the study is to assess whether the performance of type 2 quadratus lumborum block produces an improvement in the quality of life of the patient with osteoarthritis of the hip.

DETAILED DESCRIPTION:
The quadratus lumborum block is an interfascial block of the posterior wall of the abdomen, initially described for the management of postoperative pain in abdominal surgery due to its suggested effect on the T7-11 roots. The analgesic efficacy of type 1 quadratus lumborum block (QL1) in hip surgery was subsequently published. Regarding chronic pain, QL2 has been successfully performed in posttherniorrhaphy pain or pancreatic cancer.

This quadratus lumborum type 2 or posterior, is performed in the patients with hip joint based on the innervation of the hip and taking the role of thoraco-lumbar fascia in the analgesia of these patients as a reference. The good results obtained in the first 5 patients have led us to evaluate whether this blockade can indeed be an analgesic alternative in patients with coxarthrosis.

ELIGIBILITY:
Inclusion Criteria:

* Sign informed consent (Annex 2)
* Age 18-85 years
* Cartilage injury (coxarthrosis) hip
* Illness <1 year of evolution
* Patients with pain after treatment with physical therapy, exercises, NSAIDs.
* EVN> 5

Exclusion Criteria:

* Refusal of the patient
* Allergy to the drugs used
* Contraindication for performing the technique
* Intraarticular treatment in the previous 3 months
* Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient with coxalgia
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
relieve chronic hip pain | 3 months
  The main objective of the study is to assess whether the performance of type 2 lumbar .square block produces an improvement in the quality of life of the patient with osteoarthritis of the hip. The evaluation of the patient will consist of 2 stages. The first of these will consist of the evaluation consultation
  evaluation with verbal numeric scale (VNS: 0 no dolor-10 the worst pain imaginable ) if patients improve their quality of pain

SECONDARY OUTCOMES:
rate of adverse effects of the block | 3 months
  find if there is complications (hematome, kidney punction...)

OTHER OUTCOMES:
relieve chronic pain at 6 month | 6 months
  the main objective was to asses how long was the effect of the analgesia

CONTACTS AND LOCATIONS:
Overall Officials: Maria Teresa Fernandez, Study Chair — Hospital Medina del Campo
Locations (1):
- María Teresa Fernandez, Valladolid, Castille and León, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adhikary SD, Short AJ, El-Boghdadly K, Abdelmalak MJ, Chin KJ. Transmuscular quadratus lumborum versus lumbar plexus block for total hip arthroplasty: A retrospective propensity score matched cohort study. J Anaesthesiol Clin Pharmacol. 2018 Jul-Sep;34(3):372-378. doi: 10.4103/joacp.JOACP_335_17. PMID 30386022
- [Background] Adhikary SD, El-Boghdadly K, Nasralah Z, Sarwani N, Nixon AM, Chin KJ. A radiologic and anatomic assessment of injectate spread following transmuscular quadratus lumborum block in cadavers. Anaesthesia. 2017 Jan;72(1):73-79. doi: 10.1111/anae.13647. Epub 2016 Oct 12. PMID 27730633
- [Background] Fernandez Martin MT, Lopez Alvarez S, Ortigosa Solorzano E. Quadratus lumborum block. New approach for a chronic hip pain. Cases report. Rev Esp Anestesiol Reanim (Engl Ed). 2020 Jan;67(1):44-48. doi: 10.1016/j.redar.2019.10.001. Epub 2019 Nov 22. English, Spanish. PMID 31767198
- [Background] Fernandez MT, Aguirre JA, Lopez S. Posterior Quadratus Lumborum Block, A Novel Approach to Treat Chronic Hip Pain: A Case Series. A A Pract. 2023 Mar 17;17(3):e01671. doi: 10.1213/XAA.0000000000001671. eCollection 2023 Mar 1. PMID 36930793
- [Result] Fernandez Martin MT, Ortigosa E, Aguirre JA. Posterior quadratus lumborum block in chronic hip pain, preliminary results from a prospective study. Minerva Anestesiol. 2023 Mar;89(3):231-233. doi: 10.23736/S0375-9393.22.16892-6. Epub 2022 Oct 25. No abstract available. PMID 36282230